CLINICAL TRIAL: NCT06922630
Title: WIN: a Feasibility Study of a Weight-Neutral Health Intervention. Lighthouse Consortium on Obesity Management (LightCOM) Trial no 1.
Brief Title: WIN: a Feasibility Study of a Weight-Neutral Health Intervention
Acronym: WIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carsten Dirksen (Other)
Collaborators: University of Copenhagen (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Carsten Dirksen, Associate Professor, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIN feasibility study; NNF22SA0080921 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WIN (Experimental): Weight-neutral health intervention
  Interventions: Behavioral: WIN

INTERVENTIONS:
Behavioral: WIN — Weight-neutral health intervention

SUMMARY:
The WIN intervention aims to improve the mental, social and physical health as well as quality of life of participants with BMI≥30 without focusing on their weight, and with no aim of weight loss. The WIN 6 months intervention is based on the principles and methods of the weight neutral movement Health at Every Size (HAES). The content is developed in a co-design process that involved Danish participants who have lived or professional experiences with such approaches.

The intervention uses the method of intuitive eating to align eating behaviours with internal cues of hunger and fullness rather than rules, restrictions and external cues. The intervention also draws on components from Acceptance and Commitment Therapy (ACT) to manage body image concerns and weight stigma.

DETAILED DESCRIPTION:
The WIN group intervention comprises bi-weekly two-hour sessions with 11-12 participants and two WIN-therapists. Session 1 is an individual session and sessions 2-12 are group sessions. The programmes include psychoeducation, group discussions and homework about topics within the weight neutral approach such as intuitive eating, weight stigma, enjoyable movement and self-compassion.

Overview of sessions 1-12:

1. Individual session with a WIN therapist to explore the participant's expectations and needs in relation to commencing intuitive eating and body acceptance.
2. Introduction to weight-neutral health
3. Your body, Your rules
4. Intuitive eating I
5. Intuitive eating II
6. Body Respect and Weight Stigmatization
7. Self-compassion and confronting your inner critical voice
8. Body awareness, Rest and Movement - Yoga and Your strong body
9. Body awareness, Rest and Movement, intimacy and sexuality
10. Follow-up on intuitive eating
11. Follow-up on challenges
12. Strategies for resilience

Optional WIN elements include two support network events, up to 24 2-hour sessions of WIN-physical activity (Rest and Movement (12 sessions) and Competent Body Training (12 sessions)), and three individual online sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at screening.
* BMI ≥30 kg/m2.
* Residence in the Capital Region of Denmark.
* Able to understand and communicate in Danish.
* Informed consent.

Exclusion Criteria:

* Intends to become pregnant during the intervention or is currently pregnant.
* Has used weight loss medications or GLP-1 agonist treatment within the past 6 months or intends to use weight loss medications or begin any other intensive weight loss treatment during the WIN intervention.
* Has severe psychiatric or physical conditions that may interfere with participation or may present a safety concern.
* Cannot transport themselves to the group sessions.
* Is deemed unable to complete a two-hour group session, as assessed by the investigator at the clinical screening interview.
* Takes part in other research involving weight loss treatment that would compromise participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary feasibility outcome: completion of follow-up | 24 weeks after inclusion
  The proportion of participants who complete the follow-up examination, defined as answering the 'Mental health component' of the 36-item Short Form survey

SECONDARY OUTCOMES:
Secondary feasibility outcome: recruitment proportion | Inclusion
  The proportion of people who are enrolled as participants (numerator, n) out of all those who passed the initial telephone screening (denominator, N).
Secondary feasibility outcome: fidelity midway | After group session 5 (study week 12)
  Proportion of sessions attended by participants compared to the total number of sessions available
Secondary feasibility outcome: fidelity end of intervention | After group session 11 (study week 23)
  Proportion of sessions attended by participants compared to the total number of sessions available

OTHER OUTCOMES:
Exploratory feasibility outcomes: Completion of follow-up, individual questionnaires | End of study (week 24)
  Proportion of participants that complete all questionnaires required in CID1 and CID2, see list below (all outcomes specified as 'exploratory clinical outcome, questionnaire')
Exploratory feasibility outcomes: Completion of follow-up, blood samples | End of study (week 24)
  Proportion of participants willing to give blood samples at both CID1 and CID2
Exploratory feasibility outcomes: Completion of follow-up, hair samples | End of study (week 24)
  Proportion of participants willing to give hair samples at both CID1 and CID2
Exploratory feasibility outcomes: Completion of follow-up, actigraphy | End of study (week 24)
  Proportion of participants willing to wear an actigraphy measuring physical activity. Assessed as the proportion of participants willing to wear and returning the SENS monitor after both CID1 and CID2.
Exploratory feasibility outcomes: Completion of follow-up, physical assessments | End of study (week 24)
  Proportion of participants participating in the physical assessments in both CID1 and CID2, see list below (all outcomes specified as 'exploratory clinical outcome, physical assessment')
Exploratory feasibility outcomes: Compliance and participant engagement, 'rest and movement' | End of study (week 24)
  Proportion of participants participating in at least one of the optional sessions 'rest and movement'
Exploratory feasibility outcomes: Compliance and participant engagement, 'competence and strength training' | End of study (week 24)
  Proportion of participants participating in at least one of the optional sessions 'competence and strength training'
Exploratory feasibility outcomes: Compliance and participant engagement, 'support network events' | End of study (week 24)
  Proportion of participants participating in at least one of the optional 'support network events'
Exploratory feasibility outcomes: Compliance and participant engagement, 'online sessions' | End of study (week 24)
  Proportion of participants who attends at least one online session with the WIN-group therapist
Exploratory clinical outcome, questionnaire: SF-36 mental component score | End of study (week 24)
  Quality of life, Short Form 36, mental component score (scale from 0-100, higher scores indicate better mental health)
Exploratory clinical outcome, questionnaire: SF-36 physical component score | End of study (week 24)
  Quality of life, Short Form 36, physical component score (scale from 0-100, higher scores indicate better mental health)
Exploratory clinical outcome, questionnaire: SF-36 subscales | End of study (week 24)
  Quality of life, Short Form 36, individual domains (scales from 0-100, higher scores indicate better mental health):
  * physical functioning,
  * role limitations due to physical health problems,
  * bodily pain,
  * general health,
  * vitality (energy or fatigue),
  * social functioning,
  * role limitations due to emotional problems,
  * mental health (psychological distress and psychological well-being).
Exploratory clinical outcome, questionnaire: Mental health - WBIS-M | End of study (week 24)
  Weight Bias Internalization Scale (WBIS-M) score (scale from 1-7, higher scores indicate higher degree of internalized weight bias)
Exploratory clinical outcome, questionnaire: Intuitive Eating Scale - IES-3 | End of study (week 24)
  Intuitive Eating Scale measuring participants' ability to rely on internal hunger and satiety cues, reject dieting mentally, and approach eating with body respect. 12 items, each scored 1-5. Minimum value 12, maximum value 60. Higher score reflects more intuitive eating (better outcome).
Exploratory clinical outcome, questionnaire: Mental health - EDE-Q | End of study (week 24)
  Eating Disorder Examination Questionnaire (EDE-Q) score (scale from 0 to 6, higher scores indicate higher degree of eating disorder)
Exploratory clinical outcome, questionnaire: Rosenberg Self-Esteem Scale | End of study (week 24)
  Rosenberg Self-Esteem Scale, measuring self-esteem levels as a psychological marker of well-being. 10 items, each scored 1-4. Minimum value 10, maximum value 40. Higher scores indicate higher self-esteem (better outcome).
Exploratory clinical outcome, questionnaire: Body Appreciation Scale 2 | End of study (week 24)
  Body Appreciation Scale 2 (BAS-2), assessing positive body image, focusing on body acceptance and appreciation. 10 items, each scored 1-5. Minimum value 10, maximum value 50. Higher score indicates higher body appreciation (better outcome).
Exploratory clinical outcome, questionnaire: Cantril Ladder Scale | End of study (week 24)
  Cantril Ladder Scale, providing a subjective measure of life satisfaction and well-being. Range: 0-10. A ladder stretching from 0 at the bottom (worst possible situation) to 10 at the top (best possible situation). Higher score indicates a more positive evaluation of one´s life (better outcome).
Exploratory clinical outcome, questionnaire: Major Depression Inventory (MDI) | End of study (week 24)
  Major Depression Inventory (MDI) (scale from 0-50, higher scores indicate more symptoms of depression)
Exploratory clinical outcome, questionnaire: Perceived Stress Scale (PSS-10) | End of study (week 24)
  Perceived Stress Scale (PSS-10), measures perceived stress over the past month. 10 items, each scored 0-4. Minimum value 0, maximum value 40. Higher scores indicating higher perceived stress (worse outcome).
  (Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.)
Exploratory clinical outcome: physical activity, SENS | End of study (week 24)
  Assessed with activity tracker (SENS), measuring daily movement and exercise patterns (hours/day)
Exploratory clinical outcome: sleep, SENS | End of study (week 24)
  Sleep duration using SENS Motion accelerometers (hours/day)
Exploratory clinical outcome: chronic stress | End of study (week 24)
  Chronic stress (hair cortisol as a biomarker of long-term stress exposure)
Exploratory clinical outcome, physical assessment: blood pressure | End of study (week 24)
  Systolic and diastolic blood pressure (mmHg)
Exploratory clinical outcome, physical assessment: pulse | End of study (week 24)
  Pulse rate (beats per minute)
Exploratory clinical outcome, physical assessment: weight | End of study (week 24)
  Weight (kg)
Exploratory clinical outcome: Hb1Ac | End of study (week 24)
  Haemoglobin A1c (mmol/mol)
Exploratory clinical outcome: lipids | End of study (week 24)
  Lipid profile (HDL, LDL, VLDL, total cholesterol and triglycerides) (mmol/L)
Exploratory clinical outcome: creatinine | End of study (week 24)
  Creatinine (umol/L)
Exploratory clinical outcome: eGRF | End of study (week 24)
  Estimated Glomerular Filtration Rate (eGFR) (mL/min/1.73^2)
Exploratory clinical outcome: hsCRP | End of study (week 24)
  High-sensitivity C-reactive protein (hsCRP), mg/L
Exploratory clinical outcome: ALAT | End of study (week 24)
  Alanine aminotransferase (ALAT) (unit per liter)
Exploratory clinical outcome: TSH | End of study (week 24)
  Thyroid-stimulating hormone (x10^-3 IU/L)
Exploratory clinical outcome: Sodium | End of study (week 24)
  Sodium (mmol/L)
Exploratory clinical outcome: Potassium | End of study (week 24)
  Potassium (mmol/L)
Exploratory clinical outcome: Haemoglobin | End of study (week 24)
  Haemoglobin (mmol/L)
Exploratory clinical outcome: vitamin D | End of study (week 24)
  25-OH vitamin D (nmol/L)
Exploratory clinical outcome: serious adverse event | End of study (week 24)
  Proportion of participants that experienced at least one serious adverse event (according to ICH-GCP guidelines)
Other feasibility outcomes: Completion of follow-up, individual questionnaires | End of study (week 24)
  Proportion of participants that complete all questionnaires required in CID1 and CID2, see list below (all outcomes specified as 'exploratory clinical outcome, questionnaire')

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Dirksen, Ass. Professor, Study Chair — Hvidovre University Hospital
Locations (1):
- Research Unit for General Practice and Section of General Medicine, Department of Public Health, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After the results have been published, the aim is to make a depersonalised dataset publicly available on e.g. ClinicalTrials.gov and/or the European Union (EU) Zenodo database (https://zenodo.org/). The final choice will reflect which platform(s) that are compliant with current legislation at that time.
Supporting Information: Study Protocol, SAP
Time Frame: When the results have been published
Access Criteria: Researchers with a protocol for their planned study

REFERENCES:
- See also: LightCOM website — https://www.regionh.dk/lightcom/uk/Pages/default.aspx